CLINICAL TRIAL: NCT07171541
Title: Correlation Between Optical Coherence Tomography and Multifocal Electroretinogram Findings With Visual Acuity in Patients With Macular Dystrophy
Brief Title: Correlation Between OCT and Mf-ERG Findings With BCVA in Patients With Macular Dystrophy
Status: Not yet recruiting | Type: Observational
Sponsor: New Valley University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Kamel Ahmed Hassan, Dr.principle investigators/ Lecture of ophthalmology ,faculty of medicine , New Valley University, New Valley University
Other Study IDs: CBOTMEFVAPMD
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Macular Dystrophy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: OCT ,mFERG,VA test — retinal photography by OCT, VA measurement, and mfERG test

SUMMARY:
Correlation between optical coherence tomography and multifocal electroretinogram findings with visual acuity in patients with macular dystrophy.

DETAILED DESCRIPTION:
Macular dystrophies cause progressive central vision loss, but the relationship between structural retinal changes (OCT) and functional deficits (mf-ERG) with visual outcomes remains poorly understood. Current clinical assessment relies primarily on visual acuity, which inadequately reflects retinal damage or predicts disease progression. This knowledge gap limits prognostic accuracy and optimal patient management. Recent advances in OCT and mf-ERG technology provide an opportunity to establish robust structure-function correlations. Understanding these relationships will enhance patient care through improved prognosis, standardized monitoring protocols, and better clinical trial outcome measures for macular dystrophy patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with macular dystrophy in Tiba Eye Centre, Egypt, Assiut, during the period of the study

Exclusion Criteria:

* The patients diagnosed with macular dystrophy refuse to contribute to the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with macular dystrophy during the period of the study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
BCVA (best corrected visual acuity) | Day 1/month 3
  BCVA was recorded in 30 eyes of 30 patients with macular dystrophy.
CMT (central macular thickness) μm Central macular thickness measurement using optical coherence tomography | Day1/month 3
  CMT (central macular thickness) in μm in 30 eyes of 30 patients with macular dystrophy Central macular thickness measurement using optical coherence tomography.
mf-ERG amplituide nV/deg2 | Day 1/month 6
  mf-ERG amplitude nV/deg² in 30 eyes of 30 patients with macular dystrophy multifocal electroretinogram amplitude measurement using the mf-ERG machine